CLINICAL TRIAL: NCT04930900
Title: A Two-Treatment, Sequential, Crossover Study of the Pharmacokinetics of Adrenaline After Administration of ARS -1 in Subjects With Upper Respiratory Tract Infection (Infectious Rhinitis)
Brief Title: Pharmacokinetics of Adrenaline After Administration of ARS -1 in Subjects With Upper Respiratory Tract Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ARS Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EPI 014
Record Dates: First submitted 2021-06-09; First posted 2021-06-18 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Upper Respiratory Tract Infection
MeSH Terms: conditions — Respiratory Tract Infections | interventions — Cold Temperature; Epinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ARS-1 with URTI (Experimental): ARS-1 with URTI
  Interventions: Drug: ARS-1 with URTI
- ARS-1 without URTI (Experimental): ARS-1 without URTI
  Interventions: Drug: ARS-1 without URTI

INTERVENTIONS:
Drug: ARS-1 with URTI — ARS-1
  Other Names: Adrenaline
  Arms: ARS-1 with URTI
Drug: ARS-1 without URTI — ARS-1 without URTI
  Arms: ARS-1 without URTI

SUMMARY:
This is a Phase 1, single-dose, two-period study that will consist of a combined screening and baseline period and an open-label treatment period. Subjects will be enrolled when they experience an Upper Respiratory Tract Infection with nasal congestion and edema.

ELIGIBILITY:
Inclusion Criteria:

* Treatment Period 1 only, subject has symptoms of an URTI at time of dosing based on the clinical judgement and the positive infectious cause of URTI to be confirmed by Respiratory Pathogens Panel.
* Has body weight more than 55 kg for male and 50 kg for female and body mass index between 18 and 32 kg/m2, inclusive.
* Has no declared medical history of hypertension and cardiovascular disease in the last 10 years.
* At screening, has stable vital signs in the following ranges (after 5 minutes of rest):

  * SBP ≥90 and ≤140 mmHg
  * DBP ≥50 and ≤90 mmHg
  * HR ≥45 and ≤100 beats per minute (bpm)
* Is a nonsmoker within the previous 2 months (calculated from first dosing) and does not use tobacco-containing products.

Exclusion Criteria:

* Has a stated history of clinically significant gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, psychiatric, or cardiovascular disease or any other condition which, in the opinion of the Investigator, would jeopardize the safety of the subject or impact the validity of the study results.
* Has current or past history of clinically significant asthma or angioedema.
* Has prior nasal fractures, severe nasal injuries or history of nasal disorders that could interfere with nasal spray administration.
* Has any clinically significant medical condition or physical exam (PE) finding as deemed inappropriate by the Investigator.
* Has abnormal cardiovascular exam at screening including any prior history of myocardial infarction or clinically significant abnormal ECG.
* Subject reports they have had significant traumatic injury, major surgery or open biopsy within 30 days prior to study screening.
* Subject reports they have donated blood including platelets or plasma only or had an acute loss of blood (>50 mL) during the 30 days before study drug administration or intends to donate blood or blood products within 30 days after the completion of the study.
* Has a history (within 12 months before screening) of drug use, or has a positive test for drugs of abuse at screening or upon admittance to the study center, or has a stated history of alcohol abuse.
* Has been on an abnormal diet during the four (4) weeks from Day 0. 10. Has participated in a clinical trial within 30 days prior to the first dose of study drug.

  11. Has had treatment with any adrenaline or noradrenaline containing products within 7 days of Day 0.

  12. Has inadequate or difficult venous access that may jeopardize the quality or timing of the PK samples.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2021-08-09 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-07-25 (Actual)

PRIMARY OUTCOMES:
To evaluate the bioavailability (Cmax) of ARS-1 after intranasal administration | Day -1 to Day 30
  Blood samples will be collected to measure plasma concentrations of adrenaline
To evaluate the bioavailability (AUC0-t) of ARS-1 after intranasal administration | Day -1 to Day 30
  Blood samples will be collected to measure plasma concentrations of adrenaline
To evaluate the bioavailability (tmax) of ARS-1 after intranasal administration | Day -1 to Day 30
  Blood samples will be collected to measure plasma concentrations of adrenaline

CONTACTS AND LOCATIONS:
Overall Officials: Anthony McGirr, MD, Principal Investigator — Northern Beach Clinical Research Pty Ltd,
Locations (1):
- Anthony McGirr, Brookvale, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No